CLINICAL TRIAL: NCT03444038
Title: Open-Label Safety and Tolerability Study of Optimized Doses of NBI-98854 for the Treatment of Pediatric Subjects With Tourette Syndrome
Brief Title: Open-Label Safety and Tolerability Study of NBI-98854 for the Treatment of Pediatric Subjects With Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-TS2004
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-01

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valbenazine (Experimental): Valbenazine administered once daily for up to 24 weeks
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine — vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: NBI-98854

SUMMARY:
This is a Phase 2b, multicenter, open-label study to evaluate the safety and tolerability of optimized doses of NBI-98854 administered once daily for 24 weeks in pediatric subjects with Tourette Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Have participated in and completed Study NBI-98854-TS2003
2. Have a clinical diagnosis of Tourette Syndrome (TS)
3. If using maintenance medication(s) for TS or TS spectrum diagnoses (e.g. obsessive-compulsive disorder [OCD], Attention-Deficit Hyperactivity Disorder [ADHD]), be on stable doses
4. Be in good general health
5. Adolescent subjects (12 to 18 years of age) must have a negative urine drug screen for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids and a negative alcohol screen
6. Subjects of childbearing potential who do not practice total abstinence must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study

Exclusion Criteria:

1. Have an active, clinically significant unstable medical condition within 1 month prior to screening
2. Have a known history of long QT syndrome or cardiac arrhythmia
3. Have a known history of neuroleptic malignant syndrome
4. Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed)
5. Have an allergy, hypersensitivity, or intolerance to vesicular monoamine transporter 2 (VMAT2) inhibitors
6. Have a blood loss ≥250 mL or donated blood within 56 days prior to baseline
7. Have a known history of substance (drug) dependence, or substance or alcohol abuse
8. Have a significant risk of suicidal or violent behavior
9. Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (35):
- United States (34):
  - Neurocrine Clinical Site, Sun City, Arizona
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Santa Ana, California
  - Neurocrine Clinical Site, Santa Clarita, California
  - Neurocrine Clinical Site, New Haven, Connecticut
  - Neurocrine Clinical Site, Boca Raton, Florida
  - Neurocrine Clinical Site, Gulf Breeze, Florida
  - Neurocrine Clinical Site, Hialeah, Florida
  - Neurocrine Clinical Site, Orlando, Florida
  - Neurocrine Clinical Site, St. Petersburg, Florida
  - Neurocrine Clinical Site, Tampa, Florida
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Naperville, Illinois
  - Neurocrine Clinical Site, Iowa City, Iowa
  - Neurocrine Clinical Site, Leawood, Kansas
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, Bloomfield Hills, Michigan
  - Neurocrine Clinical Site, St Louis, Missouri
  - Neurocrine Clinical Site, Lincoln, Nebraska
  - Neurocrine Clinical Site, Nashua, New Hampshire
  - Neurocrine Clinical Site, Mount Arlington, New Jersey
  - Neurocrine Clinical Site, Voorhees Township, New Jersey
  - Neurocrine Clinical Site, New York, New York
  - Neurocrine Clinical Site, The Bronx, New York
  - Neurocrine Clinical Site, Durham, North Carolina
  - Neurocrine Clinical Site, Mason, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Charleston, South Carolina
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, San Antonio, Texas
  - Neurocrine Clinical Site, Everett, Washington
  - Neurocrine Clinical Site, Tacoma, Washington
- Neurocrine Clinical Site, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farber RH, Angelov A, Kim K, Carmack T, Thai-Cuarto D, Roberts E. Clinical development of valbenazine for tics associated with Tourette syndrome. Expert Rev Neurother. 2021 Apr;21(4):393-404. doi: 10.1080/14737175.2021.1898948. Epub 2021 Apr 1. PMID 33682568

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 120 male and female pediatric participants, 6 to 18 years of age, with a Diagnostic and Statistical Manual of Mental Disorders, 4th or 5th Editions (DSM-IV or -5) diagnosis of Tourette Syndrome, were planned to be enrolled. A total of 85 participants were enrolled and received at least 1 dose of study treatment.
Groups:
- Valbenazine: Participants received valbenazine once daily for up to 24 weeks. The starting dose was 20 mg for participants <50 kg at baseline and 40 mg for participants ≥50 kg at baseline, and could be escalated in increments of 20 mg every 2 weeks to a maximum of 60 mg for participants <50 kg and 80 mg for participants ≥50 kg to achieve an optimal dose of valbenazine for each participant.
Period: Overall Study
Arm/Group | Valbenazine
Started | 85
Completed | 56
Not Completed | 29
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Lack of Efficacy | 7

BASELINE CHARACTERISTICS:
Arm/Group | Valbenazine
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 3
  Race: Native Hawaiian or Other Pacific Islander | 1
  Race: Black or African American | 6
  Race: White | 72
  Race: More than one race | 0
  Race: Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is an adverse event not present prior to the initiation of study drug dosing, or is an already present event that worsens either in intensity or frequency following the initiation of study drug dosing. All qualifying TEAE are reported regardless of threshold.
Time Frame: Baseline through Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Valbenazine
Number analyzed (Participants) | 85
Participants | 71

ADVERSE EVENTS:
Time Frame: From baseline up to Week 28.
Arm/Group | Valbenazine
All-Cause Mortality (participants affected / at risk) | 0/85
Serious Adverse Events (participants affected / at risk) | 3/85
Other Adverse Events (participants affected / at risk) | 50/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine (N=85)
Infected bites (Infections and infestations) | 1
Cognitive disorder (Nervous system disorders) | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine (N=85)
Abdominal pain upper (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 11
Irritability (General disorders) | 8
Headache (Nervous system disorders) | 9
Sedation (Nervous system disorders) | 10
Somnolence (Nervous system disorders) | 17
Depression (Psychiatric disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT03444038/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT03444038/SAP_001.pdf